CLINICAL TRIAL: NCT02240914
Title: Prospective, Single-arm, Single Center, Pilot Study of Vascular Ultrasound Imaging Used as an Adjunct to Intravascular Ultrasound for Diagnosing Iliac Vein Obstruction
Brief Title: Vascular Ultrasound Versus Intravascular Ultrasound for Diagnosing Iliac Vein Obstruction
Acronym: USG-DIVO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fabio H Rossi (Other)
Collaborators: Instituto Dante Pazzanese de Cardiologia (Other); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor-Investigator, Fabio H Rossi, PHD, Instituto Dante Pazzanese de Cardiologia
Organization: Instituto Dante Pazzanese de Cardiologia (Other)
Other Study IDs: IDPC_ 4 2014
Record Dates: First submitted 2014-09-03; First posted 2014-09-16 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Iliac Vein Obstruction; May-Thurner Syndrome; Cockett Syndrome
Keywords: Iliac Vein Obstruction; May-Thurner Syndrome; Cockett Syndrome; Vascular Ultrasound; IVUS
MeSH Terms: conditions — May-Thurner Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Vascular USG and IVUS imaging diagnosis

SUMMARY:
* Determine the sensitivity, specificity and accuracy of vascular ultrasound, using direct and indirect ultrasonographic signs, in the obstructive diseases of iliac venous segment, in patients with advanced chronic venous insufficiency (CEAP 3-6), considering the intravascular ultrasound (IVUS) as the gold standard for this diagnosis.
* Develop an algorithm for noninvasive ultrasound investigation of obstructive lesions in the iliac segment in patients with advanced chronic venous insufficiency (CEAP 3-6).

ELIGIBILITY:
Inclusion Criteria:

* Advanced Chronic Venous Insufficiency (CEAP 3-6) submitted to clinical treatment for at least 1 year with no response.
* Subject must be > 18 and < 80 years of age
* Willing to participate in and able to understand, read and sign the informed consent document before the planned procedure
* On duplex ultrasound: patent common femoral vein, and patent deep femoral vein, and/or femoral vein of the study leg

Exclusion Criteria:

* Subject cannot or will not provide written informed consent
* Previous venous stent implantation involving the study leg or inferior vena cava
* Previous venovenous bypass surgery involving the study leg
* Known reaction or sensitivity to iodinated contrast that cannot be managed with premedication
* Subjects who are pregnant (women of childbearing potential must have a negative pregnancy test within 7 days prior to enrollment
* Acute deep venous thrombosis involving either leg
* Known history of chronic total occlusion of the common femoral vein of the study leg.
* Known history of thrombophilia (e.g., protein C or S deficiency, anti-thrombin III deficiency, presence of lupus anticoagulant, etc.)
* Venous compression caused by tumor encasement
* Venous outflow obstruction caused by tumor thrombus
* Life expectancy of less than 6 months
* Lower Extremity Arterial Insufficiency
* Elevated baseline blood creatinine (value greater than the upper limit of the normal range)
* Any concurrent disease or condition that, in the opinion of the Investigator, would make the subject unsuitable for participation in the study; examples include but are not limited to the inability to lie supine for the index procedure (e.g., severe congestive heart failure), thrombocytopenia or other hematological disorders associated with an unacceptable risk of bleeding, implanted orthopedic hardware that precludes proper imaging, etc.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with iliac compression disease CEAP classification 3-6.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-11 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
A composite of direct and indirect ultrasonographic signs as a measure of iliac vein stenosis | within 15 days
  • 50 patients with Clinical-Etiologic-Anatomic-Pathophysiologic (CEAP) classification C3-6 undergoing iliac and common femoral vascular ultrasound imaging with intention to detect significative iliac vein obstructions ( > 50%) and this results will be compared with the gold standard method - IVUS. Primary Endpoints: venous imaging in B- mode, volume flow and expiratory velocity in femoral vein, and the velocity relation before and through the stenosis provided by vascular ultrasound will be analyzed. Venous IVUS will provide measurements of minimum and maximum diameter reduction due to iliofemoral venous obstruction/compression; cross-sectional area reduction will also be measured.
  The percentage of significant stenosis detected at various thresholds [ < 50%, 50-80%,> 80%] with each method will be compared in a pair-wise fashion. This will be done with descriptive statistics of the detection rates for each method, and the rate of discordance between the two.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick B Metzger, MD, Principal Investigator — Vascular Surgeon
Locations (1):
- Instituto Dante Pazzanese de Cardiologia, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] MAY R, THURNER J. The cause of the predominantly sinistral occurrence of thrombosis of the pelvic veins. Angiology. 1957 Oct;8(5):419-27. doi: 10.1177/000331975700800505. No abstract available. PMID 13478912
- [Background] Cockett FB, Thomas ML. The iliac compression syndrome. Br J Surg. 1965 Oct;52(10):816-21. doi: 10.1002/bjs.1800521028. No abstract available. PMID 5828716
- [Background] Marston W, Fish D, Unger J, Keagy B. Incidence of and risk factors for iliocaval venous obstruction in patients with active or healed venous leg ulcers. J Vasc Surg. 2011 May;53(5):1303-8. doi: 10.1016/j.jvs.2010.10.120. Epub 2011 Jan 7. PMID 21215568
- [Background] Etufugh CN, Phillips TJ. Venous ulcers. Clin Dermatol. 2007 Jan-Feb;25(1):121-30. doi: 10.1016/j.clindermatol.2006.09.004. PMID 17276209
- [Background] McGuckin M, Waterman R, Brooks J, Cherry G, Porten L, Hurley S, Kerstein MD. Validation of venous leg ulcer guidelines in the United States and United Kingdom. Am J Surg. 2002 Feb;183(2):132-7. doi: 10.1016/s0002-9610(01)00856-x. PMID 11918875
- [Background] Lin EP, Bhatt S, Rubens D, Dogra VS. The importance of monophasic Doppler waveforms in the common femoral vein: a retrospective study. J Ultrasound Med. 2007 Jul;26(7):885-91. doi: 10.7863/jum.2007.26.7.885. PMID 17592051
- [Background] Neglen P, Raju S. Intravascular ultrasound scan evaluation of the obstructed vein. J Vasc Surg. 2002 Apr;35(4):694-700. doi: 10.1067/mva.2002.121127. PMID 11932665
- [Background] Labropoulos N, Borge M, Pierce K, Pappas PJ. Criteria for defining significant central vein stenosis with duplex ultrasound. J Vasc Surg. 2007 Jul;46(1):101-7. doi: 10.1016/j.jvs.2007.02.062. Epub 2007 May 30. PMID 17540535
- [Result] Virchow R. Uber die erweiterung kleiner gefasse. Arch Path Anat. 1851; 3:427.
- [Result] Malgor RD, Adrahtas D, Spentzouris G, Gasparis AP, Tassiopoulos AK, Labropoulos N. The role of duplex ultrasound in the workup of pelvic congestion syndrome. J Vasc Surg Venous Lymphat Disord. 2014 Jan;2(1):34-8. doi: 10.1016/j.jvsv.2013.06.004. Epub 2013 Sep 24. PMID 26992966
- [Result] Malgor RD, Labropoulos N. Diagnosis of venous disease with duplex ultrasound. Phlebology. 2013 Mar;28 Suppl 1:158-61. doi: 10.1177/0268355513476653. PMID 23482553
- [Result] Raju S, Hollis K, Neglen P. Obstructive lesions of the inferior vena cava: clinical features and endovenous treatment. J Vasc Surg. 2006 Oct;44(4):820-7. doi: 10.1016/j.jvs.2006.05.054. Epub 2006 Aug 22. PMID 16926084
- [Derived] Metzger PB, Rossi FH, Fernandez MG, de Carvalho SFC, Metzger SL, Izukawa NM, Kambara AM, Thorpe P. Association between the degree of iliac venous outflow obstruction by intravascular ultrasound and lower limb venous reflux. J Vasc Surg Venous Lymphat Disord. 2023 Sep;11(5):1004-1013.e1. doi: 10.1016/j.jvsv.2023.05.018. Epub 2023 Jun 21. PMID 37353155
- [Derived] Metzger PB, Rossi FH, Kambara AM, Izukawa NM, Saleh MH, Pinto IM, Amorim JE, Thorpe PE. Criteria for detecting significant chronic iliac venous obstructions with duplex ultrasound. J Vasc Surg Venous Lymphat Disord. 2016 Jan;4(1):18-27. doi: 10.1016/j.jvsv.2015.07.002. Epub 2015 Sep 12. PMID 26946891